CLINICAL TRIAL: NCT04751916
Title: Nutritional Stimulation of Muscle Protein Synthesis and Metabolic Rate After Bariatric Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oregon Health and Science University (Other)
Collaborators: The Amino Company, LLC (Unknown); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Nancy Puzziferri, Assistant Professor of Surgery, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1R44DK125151-00021210; 1R44DK125151 (NIH)
Record Dates: First submitted 2021-02-02; First posted 2021-02-12 (Actual); Last update posted 2023-04-04 (Actual); Status verified 2023-03

CONDITIONS: Weight Loss
Keywords: bariatric surgery; muscle synthesis; weight loss; essential amino acids; protein supplementation; total energy expenditure
MeSH Terms: conditions — Weight Loss

STUDY DESIGN:
Intervention Model Description: double-blinded randomized clinical trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After obtaining consent, the patient will receive supplement assignment based on computer-generated, block-randomization with stratification by sex. The intervention and control supplements are packaged, sealed and labeled as group A or B by The Amino Co. The packets are sent to Oregon Health & Science University at study start and stored at room temperature in the investigators' laboratory. The Oregon Health & Science University investigators are unaware of which supplements are packaged as group A or B. The research coordinator is responsible for completing the randomization process using a table created by the statistician. The stratification/randomization assignments are kept in a password-protected file; the password known only to the research coordinator and statistician. The powdered and reconstituted forms of the supplements are indistinguishable to an observer.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Proprietary Essential Amino Acid Protein Supplement (Experimental): Essential amino acid protein supplement; 15 grams (one packet) dissolved in 8 ounces of water twice daily for 6 months.
  Interventions: Dietary Supplement: Essential Amino Acid Protein Supplement
- Commercially-available whey protein supplement - Beneprotein® (Active Comparator): Beneprotein® whey protein supplement; 15 grams (one packet) dissolved in 8 ounces of water twice daily for 6 months.
  Interventions: Dietary Supplement: Beneprotein®

INTERVENTIONS:
Dietary Supplement: Essential Amino Acid Protein Supplement — Proprietary essential amino acid protein supplement
  Arms: Proprietary Essential Amino Acid Protein Supplement
Dietary Supplement: Beneprotein® — Whey protein supplement
  Arms: Commercially-available whey protein supplement - Beneprotein®

SUMMARY:
Bariatric surgery is an effective treatment for severe obesity but results in loss of muscle mass. The investigators will test the hypothesis that consumption of an Essential Amino Acid-based nutritional formulation will maintain muscle mass while stimulating fat loss after bariatric surgery.

DETAILED DESCRIPTION:
1. Objectives

   Bariatric surgery has become a common treatment for severe obesity, and results in a loss of fat mass. However, muscle mass is also lost following bariatric surgery. It is the investigators' overarching premise that consumption of the Essential Amino Acid-based nutritional formulation following bariatric surgery will preserve muscle mass by stimulating muscle protein synthesis. As a result, the energy utilization associated with the combination of maintained muscle mass and stimulated muscle protein synthesis will counter the decrease in metabolic rate that normally occurs in hypocaloric circumstances. Maintenance of a higher total energy expenditure by Essential Amino Acid consumption will accelerate loss of body fat, as well as accelerate loss of body weight. The investigators further propose that consumption of an Essential Amino Acid-based nutritional formulation will reduce muscle intra-cellular lipid accumulation, which will translate to greater improvements in glucose homeostasis and muscle protein metabolism. The loss of muscle mass in those with obesity undergoing rapid weight loss post-bariatric surgery, is not in itself, a disease or a medical condition.

   The following aims will test specific hypotheses related to the scientific premise:

   Aim 1. Supplementation of the usual diet following bariatric surgery with a proprietary Essential Amino Acid-based nutritional formulation twice per day for 6 months will maintain muscle mass and reduce fat mass more than supplementation of the diet with an isonitrogenous amount of whey protein. Muscle mass will be directly measured using a novel tracer-dilution technique using deuterium-labeled creatine. Fat mass and lean body mass will be measured by Dual-energy X-ray absorptiometry.

   Aim 2. Muscle protein fractional synthetic rate and total muscle protein synthesis (muscle mass x fractional synthetic rate) will decline less from pre-surgery values in participants consuming the Essential Amino Acid-based nutritional formulation as compared to whey protein. Muscle protein fractional synthetic rate will be measured by the novel "virtual biopsy" method, which provides an integrated value over three weeks.

   Aim 3. The pre-surgery rate of total energy expenditure will be better maintained in participants consuming the Essential Amino Acid-based nutritional formulation as opposed to whey protein. Change in total energy expenditure will be measured over 10-day intervals using the doubly-labeled water technique, before to 6 months following surgery.

   Aim 4. Six months after bariatric surgery muscle intra-cellular lipid accumulation will be reduced from the pre-surgery value to a greater extent in participants consuming the Essential Amino Acid-based nutritional formulation than whey protein. Muscle intra-cellular lipid accumulation will be measured by means of magnetic resonance spectroscopy and magnetic resonance imaging. The investigators anticipate that a greater reduction in intra-cellular lipid accumulation will be related to greater improvement in insulin sensitivity in terms of glucose homeostasis and also in terms of muscle protein synthesis.

   Positive results of this study will support the value of the Essential Amino Acid-based nutritional formulation in terms of increasing the rate of fat loss and improving body composition changes following bariatric surgery.
2. Background

   Despite successful weight loss and improvement of comorbidities after bariatric surgery, most patients with severe obesity remain overweight. Patients also experience variation in treatment response. Up to 30% patients experience sub-optimal weight loss or significant weight regain. Amount of weight lost and its maintenance are important because they are what lead to improvement/remission of comorbidities (diabetes, heart disease, etc.), and to decreased mortality from cardiovascular disease or cancer. One of the keys to optimal weight loss from a calorie restricted diet, and subsequent weight-loss maintenance, is losing fat without losing muscle (aka lean body mass). It is decreased energy expenditure from decreased muscle mass after weight loss which contributes significantly to weight regain. Muscle mass is the key driver of energy metabolism favoring the burning of food as fuel rather than its storage as fat. Since muscle provides a reservoir of amino acids to maintain protein synthesis essential for survival, its mass quantity is always at risk under conditions of inadequate dietary intake. Skeletal muscle, under the caloric restriction of weight-loss diets, catabolizes to provide the body's unmet protein needs. It becomes challenging to maintain muscle in conditions of severe calorie restriction such as after bariatric surgery.

   Protein supplementation has been shown to protect against muscle loss experienced in weight loss, but only if supplementation is sufficient. The standard of care approach to maintain muscle mass during rapid, significant weight loss after bariatric surgery has been dietary whey protein supplementation. After bariatric surgery, protein supplementation is limited by the inability of patients to take in sufficient calories. This can be further hindered by typical perioperative complications which limit intake, such as nausea, vomiting, and early satiety. Therefore, despite standard of care supplementation with whey protein post bariatric surgery, only marginal gains in preventing muscle loss have been made. Essential Amino Acid, the intervention supplement in this study, is a patented formula scientifically shown to be far more anabolic than whey protein in free-living elderly and young healthy adults undergoing bedrest. The Essential Amino Acid supplement stimulates protein synthesis 3-5 times as effectively as whey protein, with negligible non-protein calories.

   The importance of the role of muscle in weight loss and its maintenance cannot be overemphasized. Muscle, crucial to energy metabolism, is responsible for the majority of total energy expenditure (equivalent to physical activity energy expenditure, resting energy expenditure, and diet induced thermogenesis - calories required to digest food). Both physical activity, and muscle protein synthesis comprise a significant portion of energy expenditure. Through its function in physical activity and protein synthesis, muscle largely determines the caloric expenditure underlying the ability to 'use up' food eaten rather than store it as fat.

   Obesity, is not just increased body fat, but also increased intramuscular fat. The intramuscular fat associated with obesity impairs the muscle function of providing normal glucose homeostasis. Fortunately, when fat stored in muscle decreases, insulin sensitivity improves. Also impaired under conditions of increased intramuscular fat, is the function of providing amino acids to maintain essential protein synthesis. Impaired muscle mitochondria-stimulated protein synthesis potentially decreases resting energy expenditure, and diet induced thermogenesis. Adequate protein supplementation can counter muscle mitochondrial protein synthesis impairment, and in theory, lead to decreased intramuscular fat improving both energy expenditure and insulin sensitivity.
3. Study Design

This is a double-blinded randomized clinical trial in which the responses to consumption of one of two different dietary supplements following bariatric surgery will be determined. A variety of factors related to body composition and muscle metabolism will be quantified in participants with obesity before and approximately 6 months after bariatric surgery. This interval of time was selected because additional body weight changes are generally relatively small 6 months after surgery; most of the weight loss occurs in the first 6 months. Participants will be assigned randomly by computer to receive either an Essential Amino Acid based nutritional supplement (intervention) or a commercially-available whey protein supplement (Beneprotein®).

ELIGIBILITY:
Inclusion Criteria:

* A determination to proceed with bariatric surgery
* Roux-en-Y gastric bypass or sleeve gastrectomy
* Absence of any exclusion

Exclusion Criteria:

* Contraindications to Magnetic Resonance Spectroscopy/Magnetic Resonance Imaging
* greater than 450 pounds (scan table limit)
* Renal Failure requiring dialysis
* Liver disease as indicated by bilirubin >2 or Fibrosis-4 score ≥6
* Cardiac disease such as Left Ventricular Assist Device requirement
* Uncontrolled diabetes as indicated by Hemoglobin A1c >8
* Positive pregnancy test (for participants in whom pregnancy is possible)
* Any other exclusion per indication of clinical surgeon
* Refusal to consume study formula

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-03-09 (Actual); Primary Completion 2024-02-28 (Estimated); Study Completion 2024-02-28 (Estimated)

PRIMARY OUTCOMES:
Lean body mass | Baseline (before bariatric surgery)
  Lean body mass in kilograms
Lean body mass | 6 months after bariatric surgery
  Lean body mass in kilograms
Total energy expenditure | Baseline (before bariatric surgery)
  Total energy expenditure in kilocalories per day
Total energy expenditure | 6 months after bariatric surgery
  Total energy expenditure in kilocalories per day
Muscle mass | Baseline (before bariatric surgery)
  Muscle mass in kilograms
Muscle mass | 6 months after bariatric surgery
  Muscle mass in kilograms

SECONDARY OUTCOMES:
Liver fat mass | Baseline (before bariatric surgery)
  Liver fat mass in kilograms
Liver fat mass | 6 months after bariatric surgery
  Liver fat mass in kilograms
Visceral fat mass | Baseline (before bariatric surgery)
  Visceral fat mass in kilograms
Visceral fat mass | 6 months after bariatric surgery
  Visceral fat mass in kilograms
Subcutaneous fat mass | Baseline (before bariatric surgery)
  Subcutaneous fat mass in kilograms
Subcutaneous fat mass | 6 months after bariatric surgery
  Subcutaneous fat mass in kilograms
Whole body fat mass | Baseline (before bariatric surgery)
  Whole body fat mass in kilograms
Whole body fat mass | 6 months after bariatric surgery
  Whole body fat mass in kilograms
Weight | Baseline (before bariatric surgery)
  Weight in kilograms
Weight | 6 months after bariatric surgery
  Weight in kilograms
Resting energy expenditure | Baseline (before bariatric surgery)
  Resting energy expenditure in kilocalories per day
Resting energy expenditure | 6 months after bariatric surgery
  Resting energy expenditure in kilocalories per day
Diet induced thermogenesis | Baseline (before bariatric surgery)
  Percent kilocalories expended to digest a kilocalorie of protein
Diet induced thermogenesis | 6 months after bariatric surgery
  Percent kilocalories expended to digest a kilocalorie of protein
Glucose | Baseline (before bariatric surgery)
  Blood plasma glucose in milligrams per deciliter
Glucose | 6 months after bariatric surgery
  Blood plasma glucose in milligrams per deciliter
Insulin | Baseline (before bariatric surgery)
  Blood serum insulin in micro-international units per milliliter
Insulin | 6 months after bariatric surgery
  Blood serum insulin in micro-international units per milliliter
Essential amino acids | Baseline (before bariatric surgery)
  Blood plasma essential amino acids in micromoles per liter
Essential amino acids | 6 months after bariatric surgery
  Blood plasma essential amino acids in micromoles per liter
Dietary intake (Objective) | Baseline (before bariatric surgery)
  Dietary record of intake in kilocalories per day for 3 days
Dietary intake (Objective) | 6 months after bariatric surgery
  Dietary record of intake in kilocalories per day for 3 days
Physical activity (Objective) | Baseline (before bariatric surgery)
  Physical activity by accelerometer kilocalories per day for 7 days
Physical activity (Objective) | 6 months after bariatric surgery
  Physical activity by accelerometer kilocalories per day for 7 days
Percent muscle fat | Baseline (before bariatric surgery)
  Muscle fat in kilogram percent
Percent muscle fat | 6 months after bariatric surgery
  Muscle fat in kilogram percent
Muscle protein synthetic rate | Baseline (before bariatric surgery)
  Muscle protein synthetic rate in kilograms per day
Muscle protein synthetic rate | 6 months after bariatric surgery
  Muscle protein synthetic rate in kilograms per day
Muscle protein fractional synthetic rate | Baseline (before bariatric surgery)
  Muscle protein fractional synthetic rate in kilogram percent per day
Muscle protein fractional synthetic rate | 6 months after bariatric surgery
  Muscle protein fractional synthetic rate in kilogram percent per day

OTHER OUTCOMES:
Physical activity (Subjective) | Baseline (before bariatric surgery)
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Physical activity (Subjective) | 1 month after bariatric surgery
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Physical activity (Subjective) | 2 months after bariatric surgery
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Physical activity (Subjective) | 3 months after bariatric surgery
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Physical activity (Subjective) | 4 months after bariatric surgery
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Physical activity (Subjective) | 5 months after bariatric surgery
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Physical activity (Subjective) | 6 months after bariatric surgery
  Physical activity by self-report completion of the International Physical Activity Questionnaire
Dietary Intake (Subjective) | Baseline (before bariatric surgery)
  24-hour dietary recall collected by clinician
Dietary Intake (Subjective) | 1 month after bariatric surgery
  24-hour dietary recall collected by clinician
Dietary Intake (Subjective) | 2 months after bariatric surgery
  24-hour dietary recall collected by clinician
Dietary Intake (Subjective) | 3 months after bariatric surgery
  24-hour dietary recall collected by clinician
Dietary Intake (Subjective) | 4 months after bariatric surgery
  24-hour dietary recall collected by clinician
Dietary Intake (Subjective) | 5 months after bariatric surgery
  24-hour dietary recall collected by clinician
Dietary Intake (Subjective) | 6 months after bariatric surgery
  24-hour dietary recall collected by clinician

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Puzziferri, MD MSCS, Principal Investigator — Oregon Health and Science University
Locations (1):
- Oregon Health and Science University, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (and data dictionaries) for this study will be available once fully collected and de-identified. The study protocol, statistical analysis plan, informed consent form, and clinical study reports will also be available. Data will be available immediately following publication without an access end date. Anyone may access the data, for any purpose. Data will be available indefinitely at a link to be provided at study completion.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Immediately following publication without an access end date.
Access Criteria: Any person. Any purpose.

REFERENCES:
- [Background] Courcoulas AP, King WC, Belle SH, Berk P, Flum DR, Garcia L, Gourash W, Horlick M, Mitchell JE, Pomp A, Pories WJ, Purnell JQ, Singh A, Spaniolas K, Thirlby R, Wolfe BM, Yanovski SZ. Seven-Year Weight Trajectories and Health Outcomes in the Longitudinal Assessment of Bariatric Surgery (LABS) Study. JAMA Surg. 2018 May 1;153(5):427-434. doi: 10.1001/jamasurg.2017.5025. PMID 29214306
- [Background] Lent MR, Hu Y, Benotti PN, Petrick AT, Wood GC, Still CD, Kirchner HL. Demographic, clinical, and behavioral determinants of 7-year weight change trajectories in Roux-en-Y gastric bypass patients. Surg Obes Relat Dis. 2018 Nov;14(11):1680-1685. doi: 10.1016/j.soard.2018.07.023. Epub 2018 Jul 30. PMID 30166262
- [Background] King WC, Hinerman AS, Belle SH, Wahed AS, Courcoulas AP. Comparison of the Performance of Common Measures of Weight Regain After Bariatric Surgery for Association With Clinical Outcomes. JAMA. 2018 Oct 16;320(15):1560-1569. doi: 10.1001/jama.2018.14433. PMID 30326125
- [Background] Sjostrom L, Peltonen M, Jacobson P, Sjostrom CD, Karason K, Wedel H, Ahlin S, Anveden A, Bengtsson C, Bergmark G, Bouchard C, Carlsson B, Dahlgren S, Karlsson J, Lindroos AK, Lonroth H, Narbro K, Naslund I, Olbers T, Svensson PA, Carlsson LM. Bariatric surgery and long-term cardiovascular events. JAMA. 2012 Jan 4;307(1):56-65. doi: 10.1001/jama.2011.1914. PMID 22215166
- [Background] Adams TD, Stroup AM, Gress RE, Adams KF, Calle EE, Smith SC, Halverson RC, Simper SC, Hopkins PN, Hunt SC. Cancer incidence and mortality after gastric bypass surgery. Obesity (Silver Spring). 2009 Apr;17(4):796-802. doi: 10.1038/oby.2008.610. Epub 2009 Jan 15. PMID 19148123
- [Background] Maclean PS, Bergouignan A, Cornier MA, Jackman MR. Biology's response to dieting: the impetus for weight regain. Am J Physiol Regul Integr Comp Physiol. 2011 Sep;301(3):R581-600. doi: 10.1152/ajpregu.00755.2010. Epub 2011 Jun 15. PMID 21677272
- [Background] Leibel RL, Rosenbaum M, Hirsch J. Changes in energy expenditure resulting from altered body weight. N Engl J Med. 1995 Mar 9;332(10):621-8. doi: 10.1056/NEJM199503093321001. PMID 7632212
- [Background] Felig P, Owen OE, Wahren J, Cahill GF Jr. Amino acid metabolism during prolonged starvation. J Clin Invest. 1969 Mar;48(3):584-94. doi: 10.1172/JCI106017. PMID 5773094
- [Background] Cahill GF Jr. Starvation in man. N Engl J Med. 1970 Mar 19;282(12):668-75. doi: 10.1056/NEJM197003192821209. No abstract available. PMID 4915800
- [Background] Weijs PJM, Wolfe RR. Exploration of the protein requirement during weight loss in obese older adults. Clin Nutr. 2016 Apr;35(2):394-398. doi: 10.1016/j.clnu.2015.02.016. Epub 2015 Mar 6. PMID 25788405
- [Background] Hector AJ, McGlory C, Damas F, Mazara N, Baker SK, Phillips SM. Pronounced energy restriction with elevated protein intake results in no change in proteolysis and reductions in skeletal muscle protein synthesis that are mitigated by resistance exercise. FASEB J. 2018 Jan;32(1):265-275. doi: 10.1096/fj.201700158RR. Epub 2017 Sep 12. PMID 28899879
- [Background] Schollenberger AE, Karschin J, Meile T, Kuper MA, Konigsrainer A, Bischoff SC. Impact of protein supplementation after bariatric surgery: A randomized controlled double-blind pilot study. Nutrition. 2016 Feb;32(2):186-92. doi: 10.1016/j.nut.2015.08.005. Epub 2015 Sep 1. PMID 26691769
- [Background] Dillon EL, Sheffield-Moore M, Paddon-Jones D, Gilkison C, Sanford AP, Casperson SL, Jiang J, Chinkes DL, Urban RJ. Amino acid supplementation increases lean body mass, basal muscle protein synthesis, and insulin-like growth factor-I expression in older women. J Clin Endocrinol Metab. 2009 May;94(5):1630-7. doi: 10.1210/jc.2008-1564. Epub 2009 Feb 10. PMID 19208731
- [Background] Borsheim E, Bui QU, Tissier S, Kobayashi H, Ferrando AA, Wolfe RR. Effect of amino acid supplementation on muscle mass, strength and physical function in elderly. Clin Nutr. 2008 Apr;27(2):189-95. doi: 10.1016/j.clnu.2008.01.001. Epub 2008 Mar 4. PMID 18294740
- [Background] Paddon-Jones D, Sheffield-Moore M, Urban RJ, Sanford AP, Aarsland A, Wolfe RR, Ferrando AA. Essential amino acid and carbohydrate supplementation ameliorates muscle protein loss in humans during 28 days bedrest. J Clin Endocrinol Metab. 2004 Sep;89(9):4351-8. doi: 10.1210/jc.2003-032159. PMID 15356032
- [Background] Paddon-Jones D, Sheffield-Moore M, Katsanos CS, Zhang XJ, Wolfe RR. Differential stimulation of muscle protein synthesis in elderly humans following isocaloric ingestion of amino acids or whey protein. Exp Gerontol. 2006 Feb;41(2):215-9. doi: 10.1016/j.exger.2005.10.006. Epub 2005 Nov 23. PMID 16310330
- [Background] Kim IY, Park S, Smeets ETHC, Schutzler S, Azhar G, Wei JY, Ferrando AA, Wolfe RR. Consumption of a Specially-Formulated Mixture of Essential Amino Acids Promotes Gain in Whole-Body Protein to a Greater Extent than a Complete Meal Replacement in Older Women with Heart Failure. Nutrients. 2019 Jun 17;11(6):1360. doi: 10.3390/nu11061360. PMID 31212940
- [Background] Katsanos CS, Kobayashi H, Sheffield-Moore M, Aarsland A, Wolfe RR. A high proportion of leucine is required for optimal stimulation of the rate of muscle protein synthesis by essential amino acids in the elderly. Am J Physiol Endocrinol Metab. 2006 Aug;291(2):E381-7. doi: 10.1152/ajpendo.00488.2005. Epub 2006 Feb 28. PMID 16507602
- [Background] Goodpaster BH, Theriault R, Watkins SC, Kelley DE. Intramuscular lipid content is increased in obesity and decreased by weight loss. Metabolism. 2000 Apr;49(4):467-72. doi: 10.1016/s0026-0495(00)80010-4. PMID 10778870
- [Background] Goodpaster BH, Thaete FL, Kelley DE. Thigh adipose tissue distribution is associated with insulin resistance in obesity and in type 2 diabetes mellitus. Am J Clin Nutr. 2000 Apr;71(4):885-92. doi: 10.1093/ajcn/71.4.885. PMID 10731493
- [Background] Petersen KF, Shulman GI. Pathogenesis of skeletal muscle insulin resistance in type 2 diabetes mellitus. Am J Cardiol. 2002 Sep 5;90(5A):11G-18G. doi: 10.1016/s0002-9149(02)02554-7. PMID 12231074
- [Background] Guillet C, Delcourt I, Rance M, Giraudet C, Walrand S, Bedu M, Duche P, Boirie Y. Changes in basal and insulin and amino acid response of whole body and skeletal muscle proteins in obese men. J Clin Endocrinol Metab. 2009 Aug;94(8):3044-50. doi: 10.1210/jc.2008-2216. Epub 2009 May 26. PMID 19470633
- [Background] Liang C, Curry BJ, Brown PL, Zemel MB. Leucine Modulates Mitochondrial Biogenesis and SIRT1-AMPK Signaling in C2C12 Myotubes. J Nutr Metab. 2014;2014:239750. doi: 10.1155/2014/239750. Epub 2014 Oct 7. PMID 25400942
- [Background] Bohe J, Low JF, Wolfe RR, Rennie MJ. Latency and duration of stimulation of human muscle protein synthesis during continuous infusion of amino acids. J Physiol. 2001 Apr 15;532(Pt 2):575-9. doi: 10.1111/j.1469-7793.2001.0575f.x. PMID 11306673